CLINICAL TRIAL: NCT05318651
Title: Determinants of Use of Mobile Apps for Smoking Cessation
Brief Title: Use Determinants of Smoking Cessation App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paris Nanterre University (Other)
Responsible Party: Principal Investigator, Luz BUSTAMANTE, Principal Investigator, Paris Nanterre University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A20273336
Record Dates: First submitted 2022-03-09; First posted 2022-04-08 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Smoking Cessation; Technology Acceptance Model; CBT; Engagement
Keywords: E health; smoking cessation; engagement determinants; intention to use; TAM model
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mobile app users (Experimental)
  Interventions: Device: Kwit SAS - smoking cessation app

INTERVENTIONS:
Device: Kwit SAS - smoking cessation app — Kwit is a mobile app for smoking cessation. Different CBT techniques are used by the app already been proved as effective : Case analysis craving tool, Achievements badges,Diary, Goal (outcome) setting, A 9-steps preparation program, psychological education, Emotional monitoring, Access to groups on social networks, different strategies ( NRT/water/meditation), Motivational cards.

SUMMARY:
The development of mobile applications ("mobile apps") is steadily increasing and appears to be a promising treatment method to help people change unwanted behaviors or maintain a regular relationship with the medical system. Mobile apps aimed at smoking cessation have been shown to be effective. However, if a treatment is not used regularly, it will not have the desired effect. The main objective of this study is to identify what makes a person decide to use a smoking cessation app and to do so regularly. The second objective is to determine what is necessary to achieve long-term change with a mobile app.

DETAILED DESCRIPTION:
Despite the significant decrease in tobacco consumption in France (30% in 2000 vs. 25.4% in 2018), the prevalence of smokers aged 18 to 75 years is still a public issue. Among the new solutions proposed, mobile applications ("mobile apps") seem to be a promising treatment modality. Several advantages to their use are recognized for patients, health professionals and the health system itself. Mobile applications allow accessibility to care and information, the possibility of transposing several proven effective therapeutic principles, the possibility of integrating certain forms of information transmission such as messaging, behavioural feedback and audiovisual media.

Although mobile app development is a growing market, knowledge about the determinants of intention to use this type of technology is very limited, especially for smoking cessation apps. The investigators propose a theoretical model to examine what determines the regular use of mobile apps for smoking cessation among those who want to quit. The investigators use the TAMII model and the operational variables used in a more general study on e-health applications. A chronological organisation based on a three-part behavioural model (antecedent, target behaviour and outcome) is added to the TAMII model. The main objective is to identify the factors of Mobila App Sustain Use (MASU). All definitions of TAM-II will be used : perceived usefulness (PU), perceived ease of use (PEOU) and social norm (SN), as well as the definitions proposed by Choi et al (2014) on the predictors of PU, PEOU and SN.

ELIGIBILITY:
Participants must meet four inclusion criteria for the study:

Inclusion criteria

* Age: Be 18 years of age or older,
* Smoking Status: consider themselves an active smoker
* Motivation to quit: be willing to quit smoking, in the short and medium term.
* Agreement to participate: They must also agree to participate in the study. They will have read the information note where the procedure is described; the researchers presented and their rights to withdraw from the study are recalled.

Exclusion criteria:

* Participants must have a smartphone with an iOS or Android operating system
* Access to the internet to complete the questionnaires
* Download the application and receive the updates it offers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
First Use | Day 1 - First use
  The ratio of people accessing the app after giving them access to it.
Mobile App Sustain Use (MASU) | 90 days post firs use of the mobile apps
  The ratio of times the application is accessed per week..
Mobile App Intention Use (MAIU): | Day 15
  Questionaire : please specify by selecting a number from 1 to 3, with 1 being "Just once", 2 being "Daily" and 3 being "Several times a day", how often you expect to use this application in the course of :
  1. In the next week
  2. In the next month
Mobile App Intention Use (MAIU): | Day 30
  Questionaire : please specify by selecting a number from 1 to 3, with 1 being "Just once", 2 being "Daily" and 3 being "Several times a day", how often you expect to use this application in the course of :
  1. In the next week
  2. In the next month
Mobile App Intention Use (MAIU): | Day 60
  Questionaire : please specify by selecting a number from 1 to 3, with 1 being "Just once", 2 being "Daily" and 3 being "Several times a day", how often you expect to use this application in the course of :
  1. In the next 15 days
  2. In the next month
Mobile App Intention Use (MAIU): | Day 90
  Questionaire : Please specify by selecting a number from 1 to 3, with 1 being "Just once", 2 being "Daily" and 3 being "Several times a day", how often you expect to use this application in the course of :
  1. In the next week
  2. In the next month
Mobile App Satisfaction assessment (MAS): | Day 15
  The Mobile App Ratting Scale (MARS) scale is a multidimensional metric that ranks and assesses the quality of mobile apps. The MARS total score can be used to evaluate and compare the quality of an application with others. The total score is calculated as the average of its five categories: user engagement, functionality, aesthetics, information and subjective quality. Each category is rated on a five-point scale ranging from inadequate-1 to excellent-5 (25).This scale has been used previously to assess the quality of smoking cessation apps in the Australian market with high inter-rater reliability (ICC =0.807)
Mobile App Satisfaction assessment (MAS): | Day 30
  The Mobile App Ratting Scale (MARS) scale is a multidimensional metric that ranks and assesses the quality of mobile apps. The MARS total score can be used to evaluate and compare the quality of an application with others. The total score is calculated as the average of its five categories: user engagement, functionality, aesthetics, information and subjective quality. Each category is rated on a five-point scale ranging from inadequate-1 to excellent-5 (25).This scale has been used previously to assess the quality of smoking cessation apps in the Australian market with high inter-rater reliability (ICC =0.807)
Mobile App Satisfaction assessment (MAS): | Day 60
  The Mobile App Ratting Scale (MARS) scale is a multidimensional metric that ranks and assesses the quality of mobile apps. The MARS total score can be used to evaluate and compare the quality of an application with others. The total score is calculated as the average of its five categories: user engagement, functionality, aesthetics, information and subjective quality. Each category is rated on a five-point scale ranging from inadequate-1 to excellent-5 (25).This scale has been used previously to assess the quality of smoking cessation apps in the Australian market with high inter-rater reliability (ICC =0.807)
Mobile App Satisfaction assessment (MAS): | Day 90
  The Mobile App Ratting Scale (MARS) scale is a multidimensional metric that ranks and assesses the quality of mobile apps. The MARS total score can be used to evaluate and compare the quality of an application with others. The total score is calculated as the average of its five categories: user engagement, functionality, aesthetics, information and subjective quality. Each category is rated on a five-point scale ranging from inadequate-1 to excellent-5.This scale has been used previously to assess the quality of smoking cessation apps in the Australian market with high inter-rater reliability (ICC =0.807).

SECONDARY OUTCOMES:
Smoking profile (SP) | 1 day before the first use of the mobile app
  The degree of dependence is assessed by the Fagerström Test, which is widely used.
Craving intensity (CI) | 1 day before before the first use of the mobile app
  The visual analog scale or VAS was used to measure the average craving intensity .
Craving intensity (CI) | Day 15
  The visual analog scale or VAS was used to measure the average craving intensity .
Craving intensity (CI) | Day 30
  The visual analog scale or VAS was used to measure the average craving intensity .
Craving intensity (CI) | Day 60
  The visual analog scale or VAS was used to measure the average craving intensity .
Craving intensity (CI) | Day 90
  The visual analog scale or VAS was used to measure the average craving intensity .
Behavior change : Smoking cessation | Day 15
  Self-reported 15-day point prevalence smoking status. Since your first use of the app have you smoked a cigarette (even a puff)?
Behavior change : Smoking cessation | Day 30
  Self-reported 30-day point prevalence smoking status. Since your first use of the app have you smoked a cigarette (even a puff)?
Behavior change : Smoking cessation | Day 60
  Self-reported 60-day point prevalence smoking status. Since your first use of the app have you smoked a cigarette (even a puff)?
Behavior change : Smoking cessation | Day 90
  Self-reported 90-day point prevalence smoking status. Since your first use of the app have you smoked a cigarette (even a puff)?

CONTACTS AND LOCATIONS:
Overall Officials: Lucia ROMO, Principal Investigator — Pr. de psychologie clinique UNIVERSITE PARIS NANTERRE
Locations (1):
- Universite Paris Nanterre, Epscp, La Defense, Nanterre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor GMJ, Dalili MN, Semwal M, Civljak M, Sheikh A, Car J. Internet-based interventions for smoking cessation. Cochrane Database Syst Rev. 2017 Sep 4;9(9):CD007078. doi: 10.1002/14651858.CD007078.pub5. PMID 28869775
- [Background] Whittaker R, McRobbie H, Bullen C, Rodgers A, Gu Y. Mobile phone-based interventions for smoking cessation. Cochrane Database Syst Rev. 2016 Apr 10;4(4):CD006611. doi: 10.1002/14651858.CD006611.pub4. PMID 27060875
- [Background] Whittaker R, McRobbie H, Bullen C, Rodgers A, Gu Y, Dobson R. Mobile phone text messaging and app-based interventions for smoking cessation. Cochrane Database Syst Rev. 2019 Oct 22;10(10):CD006611. doi: 10.1002/14651858.CD006611.pub5. PMID 31638271
- [Background] Regmi K, Kassim N, Ahmad N, Tuah NA. Effectiveness of Mobile Apps for Smoking Cessation: A Review. Tob Prev Cessat. 2017 Apr 12;3:12. doi: 10.18332/tpc/70088. eCollection 2017. PMID 32432186
- [Background] Hoeppner BB, Hoeppner SS, Seaboyer L, Schick MR, Wu GW, Bergman BG, Kelly JF. How Smart are Smartphone Apps for Smoking Cessation? A Content Analysis. Nicotine Tob Res. 2016 May;18(5):1025-31. doi: 10.1093/ntr/ntv117. Epub 2015 Jun 4. PMID 26045249
- [Background] Rajani NB, Weth D, Mastellos N, Filippidis FT. Adherence of popular smoking cessation mobile applications to evidence-based guidelines. BMC Public Health. 2019 Jun 13;19(1):743. doi: 10.1186/s12889-019-7084-7. PMID 31196062
- [Background] Cho J, Quinlan MM, Park D, Noh GY. Determinants of adoption of smartphone health apps among college students. Am J Health Behav. 2014 Nov;38(6):860-70. doi: 10.5993/AJHB.38.6.8. PMID 25207512
- [Background] Cotten SR, Gupta SS. Characteristics of online and offline health information seekers and factors that discriminate between them. Soc Sci Med. 2004 Nov;59(9):1795-806. doi: 10.1016/j.socscimed.2004.02.020. PMID 15312915
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Zelenko O, Tjondronegoro D, Mani M. Mobile app rating scale: a new tool for assessing the quality of health mobile apps. JMIR Mhealth Uhealth. 2015 Mar 11;3(1):e27. doi: 10.2196/mhealth.3422. PMID 25760773
- [Background] Rajani NB, Mastellos N, Filippidis FT. Self-Efficacy and Motivation to Quit of Smokers Seeking to Quit: Quantitative Assessment of Smoking Cessation Mobile Apps. JMIR Mhealth Uhealth. 2021 Apr 30;9(4):e25030. doi: 10.2196/25030. PMID 33929336
- [Background] Rahimi B, Nadri H, Lotfnezhad Afshar H, Timpka T. A Systematic Review of the Technology Acceptance Model in Health Informatics. Appl Clin Inform. 2018 Jul;9(3):604-634. doi: 10.1055/s-0038-1668091. Epub 2018 Aug 15. PMID 30112741